CLINICAL TRIAL: NCT00150306
Title: A Multicenter, 10-Week, Randomized, Double-Blind Study Of Sertraline And Placebo In Children And Adolescents With Posttraumatic Stress Disorder (PTSD)
Brief Title: A Ten-Week Study Evaluating The Effectiveness And Safety Of Zoloft In Children And Adolescents With A Diagnosis Of PTSD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Please see Detailed Description below for termination reason.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0501061
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Zoloft (Sertraline)

SUMMARY:
To evaluate the safety and efficacy of sertraline compared to placebo in children and adolescents (6 to 17 years of age) who are outpatients with Posttraumatic Stress Disorder.

DETAILED DESCRIPTION:
This study was terminated on July 11, 2007. The results of the primary endpoint analysis at the interim showed that the Zoloft group was not significantly different than the placebo on the primary endpoint and therefore the decision was made to terminate the trial. The decision to terminate the trial was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be from 6 to 17 years of age and will have a maximum age of 17 at the Baseline Visit of the study.
* Subjects must have a diagnosis of Posttraumatic Stress Disorder as defined by DSM-IV and determined by the Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL).

Exclusion Criteria:

* Subjects whose trauma is ongoing, or who are living in the same home as their abuser, or who are expected to participate in litigation related to their trauma during the course of the study will be excluded from participation.
* Subjects who are likely to or are at high risk for experiencing re-exposure to their index trauma.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160
Dates: Start 2002-11; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The primary efficacy parameter is the University of California at Los Angeles Post-Traumatic Stress Disorder Index for DSM-IV (UCLA PTSD-I).

SECONDARY OUTCOMES:
Secondary efficacy measures include
Child Stress Disorder Checklist (CSDC)
Clinical Global Impression Severity (CGI-S)
Clinical Global Impression Improvement (CGI-I)
Children's Depression Rating Scale - Revised edition (CDRS-R)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- United States (23):
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Marcos, California
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Terre Haute, Indiana
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Bethesda, Maryland
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, Manhasset, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Stony Brook, New York
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Lyndhurst, Ohio
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Galveston, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Plano, Texas

REFERENCES:
- [Derived] Robb AS, Cueva JE, Sporn J, Yang R, Vanderburg DG. Sertraline treatment of children and adolescents with posttraumatic stress disorder: a double-blind, placebo-controlled trial. J Child Adolesc Psychopharmacol. 2010 Dec;20(6):463-71. doi: 10.1089/cap.2009.0115. PMID 21186964
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0501061&StudyName=A%20Ten-Week%20Study%20Evaluating%20The%20Effectiveness%20And%20Safety%20Of%20Zoloft%20In%20Children%20And%20Adolescents%20With%20A%20Diagnosis%20Of%20PTSD